CLINICAL TRIAL: NCT06114446
Title: The Evaluation of the Effectiveness of Colorectal Surgery Nursing Care Education Given to Nursing Students Via an Immersive Virtual Reality Environment
Brief Title: The Evaluation of the Effectiveness of Nursing Care Education Provided With Immersive Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Elif Akyüz, Principal Investigator, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EAkyuz
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Virtual Reality; Nursing Care; Colorectal Surgery; Nursing Student; Education
Keywords: colorectal surgery; education technologies; nursing education; immersive virtual reality; nursing students; nursing care
MeSH Terms: interventions — Observation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will be educated with immersive virtual reality simulation for postoperative nursing care of a patient who underwent colorectal surgery
  Interventions: Other: immersive virtual reality; Other: observation
- Control group (Other): Participants will be educated with simulation manikin for postoperative nursing care of a patient who underwent colorectal surgery
  Interventions: Other: simulation group; Other: observation

INTERVENTIONS:
Other: simulation group — Participants will be educated with simulation manikin for postoperative nursing care of a patient who underwent colorectal surgery
  Arms: Control group
Other: immersive virtual reality — Participants will be educated with immersive virtual simulation f for postoperative nursing care of a patient who underwent colorectal surgery
  Arms: Experimental group
Other: observation — All participants who participate in simulation or immersive virtual arms will be observed to assess postoperative nursing care skills

SUMMARY:
Nursing education is composed of both theoretical and practical training that complement each other. The clinical practice environment for students is quite complex and practical applications are highly variable. Practical application areas do not offer effective and equal opportunities to meet the learning and application goals. There are also problems in theoretical education, and current teaching techniques cannot adequately support students' learning. In nursing education, it is recommended to use different teaching methods that strengthen students' skills. One of these methods is virtual reality simulation, which simulates real-life procedures.

The investigators's aim in this project is to reveal the effect of the use of immersive virtual reality on the effectiveness of education in surgical nursing education through nursing care offered for a specific surgical procedure. With the laboratory setup, software tool(s), and the self-sufficient employees being able to use the software, via the capabilities gained through this project, it will be possible to carry out various types of virtual reality training activities by different departments of investigator's university without the need for out-sourcing. The investigators's advanced goal in this project is to transfer the nursing care specific to frequently applied surgical interventions to the immersive virtual reality environment.

DETAILED DESCRIPTION:
This study uses the randomized controlled experiment method with pretest-posttest. The population of the study is the students taking surgical disease care courses (100-110 students per year). The required sample size was calculated by reviewing similar studies in the literature and using the G * Power 3.1 program. It was decided that the sample would consist of 35 experimental and 35 control groups. The data collection forms (knowledge level, observed skills, and self-evaluation of clinical skill competence) were developed by the researchers based on the literature.

In this study, there are 2 groups, experimental and control groups, and at the end of the study, investigators will observe all group members individually.

At the beginning of the study, data collection forms will be completed in all groups. All participants will be asked to perform ostomy care on standardized patients. During this time, students' nursing skills will be observed individually.

Colorectal surgery nursing care will be performed in an immersive virtual reality environment in the experimental group and on a practice manikin in the nursing skills laboratory in the control group. Participants in both the control and the virtual reality groups will be included in the debriefing. After the implementation participants will complete the data collection forms again. All participants will be asked to perform ostomy care on standardized patients. During this time, students' nursing skills will be observed individually.

The quantitative data to be obtained will be analyzed using Statistical Package for Social Science (SPSS).

The simulation scenario, which will be transferred to an immersive virtual environment, includes early and late postoperative care of a patient who underwent colorectal surgery.

The research will begin in the second semester of the 2023-2024 academic year in the surgical nursing course after the completion of the data collection tools and will be completed in one academic year.

ELIGIBILITY:
Inclusion Criteria:

* to be a second-grade student
* to be taking the Surgical Diseases Nursing course,

Exclusion Criteria:

* to have taken the course before
* to repeat the course
* enter the semester through vertical or horizontal transfer programs
* graduate of a vocational high school

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Colorectal Surgery Nursing Care Knowledge Assessment Form | one day
  Investigators will use a form to measure participants' knowledge level related to colorectal surgery care. The form includes 20 questions and will be used it several times (before the implementation, two times after the implementation). Evaluation will be made out of 100 points. Higher scores will mean a better outcome.
Ostomy Care Skills Observation Form | one day
  Investigators will use a checklist to determine the participants's nursing care skills. Investigators will observe all participants during nursing care with standardized patient. The checklist includes 20 nursing care skills related to ostomy care and will be used before and after the implementation. Evaluation will be made out of 100 points. Higher scores will mean a better outcome.
Participant's Clinical Skill Competence Self Evaluation Form | one day
  This form will be used for participants's self-evaluation of skill competence. This form consists of 20 nursing care skills related to postoperative colorectal surgery patient care. It will be used before and after the implementation. Evaluation will be made out of 100 points. Higher scores will mean a better outcome.

SECONDARY OUTCOMES:
Participants' experiences of immersive virtual reality | one day
  This form will be used for getting participants' virtual reality experiences and opinions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No